CLINICAL TRIAL: NCT02502019
Title: Prospective, Multicenter, Single-arm Pilot Clinical Investigation Evaluating the Use of a Surface Bleeding Severity Scale (SBSS) and the Safety and Efficacy of a New Hemostatic Device in Abdominal and Orthopedic Lower Extremity Surgeries
Brief Title: HEMOBLAST Pilot Clinical Investigation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC 2015-001
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HEMOBLAST (Experimental): All subjects will have the investigational device implanted
  Interventions: Device: HEMOBLAST Bellows

INTERVENTIONS:
Device: HEMOBLAST Bellows — HEMOBLAST™ Bellows is intended for use in surgical procedures as an adjunct to hemostasis when control of bleeding by conventional procedures is ineffective or impractical.

SUMMARY:
The primary objective of this pilot clinical investigation is to assess the reliability of the Surface Bleeding Severity Scale (SBSS) in a clinical setting. Secondary objectives of this clinical investigation are to collect initial data on the safety and efficacy of HEMOBLAST™ Bellows in abdominal and orthopedic lower extremity surgeries.

DETAILED DESCRIPTION:
HEMOBLAST™ Bellows is intended for use in surgical procedures as an adjunct to hemostasis when control of bleeding by conventional procedures is ineffective or impractical.

This is a prospective, multicenter, single-arm pilot clinical investigation. There will be 36 subjects enrolled across 4 investigational sites.

The subjects will be followed at hospital charge and 6 weeks postoperatively.

The primary endpoint of this clinical investigation is the mean paired Kappa statistic for the assignment of SBSS scores by 2 Investigators.

Secondary endpoints of this clinical investigation consist of:

* Proportion of subjects achieving hemostasis within 6 minutes of HEMOBLAST™ Bellows application;
* Proportion of subjects achieving hemostasis within 10 minutes of HEMOBLAST™ Bellows application;
* Proportion of subjects achieving hemostasis within 3 minutes of HEMOBLAST™ Bellows application; and
* Incidence of adverse events through final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is undergoing an elective open abdominal or orthopedic lower extremity surgery;

  * Subject or an authorized legal representative is willing and able to give prior written informed consent for investigation participation;
  * Subjects on antiplatelets, including aspirin, will discontinue medication at least 10 days prior to surgery; and
  * Subject is 21 years of age or older.
  * Subject does not have an active or suspected infection at the surgical site;
  * Subject in whom the Investigator is able to identify a target bleeding site (TBS) for which any applicable conventional means for achieving hemostasis are ineffective or impractical; and
  * Subject has a TBS with an SBSS score of 1, 2, or 3.

Exclusion Criteria:

* • Subject is undergoing a laparoscopic, thoracoscopic, or robotic surgical procedure;

  * Subject is undergoing a spinal surgical procedure;
  * Subject is undergoing a neurologic surgical procedure;
  * Subject is undergoing an emergency surgical procedure;
  * Subject is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding;
  * Subject has a clinically significant coagulation disorder or disease, defined as a platelet count < 100,000 per microliter and/or International Normalized Ratio > 1.5 within 4 weeks of surgery;
  * Subject had chronic corticosteroid use within 2 weeks prior to surgery;
  * Subject receiving intravenous heparin or oral Coumadin within 24 hours of surgery;
  * Subject has an active or suspected infection at the surgical site;
  * Subject has had or has planned any organ transplantation;
  * Subject has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
  * Subject has ASA classification of > 4;
  * Subject has a life expectancy of less than 3 months;
  * Subject has a known psychiatric disorder, which in the opinion of the Principal Investigator, would preclude the subject from completing this clinical study;
  * Subject has a documented severe congenital or acquired immunodeficiency;
  * Subject has religious or other objections to porcine or bovine components;
  * Subject in whom the investigational device will be used at the site of a cemented or uncemented porous coated joint implant;
  * Subject is currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent; and
  * Subject is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Sher, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Danville Orthopedic Clinic, Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- HEMOBLAST: Subjects received the investigational device, HEMOBLAST Bellows.
Period: Overall Study
Arm/Group | HEMOBLAST
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Paired Kappa Statistic for the Assignment of SBSS Scores by 2 Investigators
Description: The primary endpoint of this clinical investigation is the mean paired Kappa statistic for the assignment of SBSS scores by 2 Investigators.
Time Frame: Intraoperative
Measure: Number; unit: Kappa statistic
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 27
Kappa statistic | 0.7754

2. Secondary Outcome: Hemostatic Within 6 Minutes
Description: Proportion of subjects achieving hemostasis within 6 minutes of HEMOBLAST™ Bellows application
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 24
Participants | 19

3. Secondary Outcome: Hemostasis Within 10 Minutes
Description: Proportion of subjects achieving hemostasis within 10 minutes of HEMOBLAST™ Bellows application
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 24
Participants | 22

4. Secondary Outcome: Hemostasis Within 3 Minutes
Description: Proportion of subjects achieving hemostasis within 3 minutes of HEMOBLAST™ Bellows application
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 24
Participants | 12

5. Secondary Outcome: Adverse Events
Description: Incidence of adverse events through final follow-up
Time Frame: 6 +/- 2 weeks after implant
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST
Number analyzed (Participants) | 27
Participants | 15

ADVERSE EVENTS:
Arm/Group | HEMOBLAST
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEMOBLAST (N=27)
Metabolic encephalopathy (General disorders) | 1 (1)
Non-occlusive thrombus and nonresponsiveness (General disorders) | 1 (1)
Pancreatic leak (Hepatobiliary disorders) | 1 (1)
Syncopy (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEMOBLAST (N=27)
Non-serious AE (General disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No